CLINICAL TRIAL: NCT04155216
Title: A Guided Meditation Program in Patients Undergoing Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1706018340
Record Dates: First submitted 2019-02-11; First posted 2019-11-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided imagery (Experimental): Relaxation and guided imagery program
  Interventions: Behavioral: Relaxation and guided imagery program

INTERVENTIONS:
Behavioral: Relaxation and guided imagery program — Listening to a relaxation and guided imagery program for 25 minutes during hemodialysis treatments.

SUMMARY:
This is an open-label, single center, non-randomized, single-arm pilot study to determine the ability of a Relaxation and Guided Imagery Program for its ability to induce a reduction in anxiety in subjects undergoing hemodialysis for End Stage Renal Disease (ESRD). Measures will evaluate the program's ability to impact anxiety, with secondary analysis of headaches, insomnia, fatigue, and pain. Subjects will be administered questionnaires at the study start and study end. Intervention will involve listening to a pre-recorded guided relaxation and imagery during regularly-scheduled dialysis sessions for four weeks.

DETAILED DESCRIPTION:
The investigators hypothesize that participation in the guided relaxation and imagery sessions, at least once during each hemodialysis session by subjects presenting with anxiety, will result in a demonstrated ability to shift out of anxiety into a peaceful state of mind, and result in a decrease in the reported immediate and overall anxiety levels.

Intervention will involve listening to a pre-recorded guided relaxation and imagery during regularly-scheduled dialysis sessions for four weeks. Subjects will be asked to complete the Kidney Disease and Quality of Life (KDQOL) questionnaire relating to quality of life measures, Likert scales to measure anxiety, headaches, insomnia, fatigue and pain and a questionnaire to assess other practiced meditative therapies, psychological therapies and medications.

Study Procedures:

Baseline: Following consent, each subject will be given an introduction to the program and will be provided with an MP3 player, pre-loaded with a recording of the guided mediation program. Subjects will be asked to complete the KDQOL questionnaire, as well as a Likert Scale to measure the psychophysical parameters in question at baseline. Subjects will be given a short questionnaire to assess other practiced meditative therapies. Per standard of care, patients will have blood drawn to measure C Reactive Protein (CRP) levels on day of consent, or within one week prior to Visit 1.

Visits 1 - 12: Subjects will complete a Likert Scale at the start of every dialysis session for 4 weeks (a total of 12 sessions), as well as listen to the recording at least once during each of the 12 sessions. Every recorded session will last approximately 25 minutes. Subjects will repeat the Likert Scale completion following each recorded session.

Visit 12: Subjects will be asked to complete the KDQOL questionnaire and a short questionnaire to assess other practiced meditative therapies, psychological therapies, and medications. Subjects will have C reactive protein drawn as standard of care. The subject's medical record will be reviewed for data relevant to the study. This includes dialysis attendance, notes on study measures, including anxiety, as well as headaches, insomnia, fatigue, and pain, KDQOL results, and CRP levels.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females; 18 years or older.
2. Receiving hemodialysis at The Rogosin Institute for End Stage Renal Disease.
3. Willingness to adhere to the treatment intervention schedule.
4. Subjects must present with anxiety.
5. Willing and able to provide informed consent.

Exclusion Criteria:

1. Plans to withdraw from dialysis at The Rogosin Institute within the study timeline.
2. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life Score | Four weeks
  To determine the quality of life using the Kidney Disease and Quality of Life (KDQOL) questionnaire. The score is determined by transforming the raw precoded numeric values of items to a 0-100 possible range, with higher transformed scores always reflecting better quality of life. Each item is put on a 0-100 range so that the lowest and highest possible score are set at 0 and 100 respectively. Scores represent the percentage of total possible score achieved.
Anxiety level | Four weeks
  To determine how much of an impact anxiety had on the subject's day to day life, using a Likert Scale, ranging from 1 (none) to 5 (extreme).

SECONDARY OUTCOMES:
Inflammation level | Four weeks
  CRP laboratory test
Headaches | Four weeks
  To determine how much of an impact headaches had on the subject's day to day life, using a Likert Scale, ranging from 1 (none) to 5 (extreme).
Insomnia | Four weeks
  To determine how much of an impact insomnia had on the subject's day to day life, using a Likert Scale, ranging from 1 (none) to 5 (extreme).
Fatigue | Four weeks
  To determine how much of an impact fatigue had on the subject's day to day life, using a Likert Scale, ranging from 1 (none) to 5 (extreme).
Feeling pain | Four weeks
  To determine how much of an impact pain had on the subject's day to day life, using a Likert Scale, ranging from 1 (none) to 5 (extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bohmart, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No